CLINICAL TRIAL: NCT01535690
Title: Photodynamic Therapy Associated With Full-mouth Ultrasonic Debridement in the Treatment of Severe Chronic Periodontitis: a Randomized-controlled Clinical Trial Running Title: Photodynamic Therapy Associated With Periodontal Debridement
Brief Title: Photodynamic Therapy Associated With Full-mouth Ultrasonic Debridement in the Treatment of Severe Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Principal Investigator, Maybel Lages Balata, Master, Escola Bahiana de Medicina e Saude Publica
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PDTMLB
Record Dates: First submitted 2012-02-04; First posted 2012-02-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Periodontitis
Keywords: Laser; Clinical trial; Non-surgical periodontal therapy; Periodontitis; bleeding on probing and radiographic bone loss; minimum of 2 teeth with probing depth (PD) ≥ 7 mm and; 2 other teeth with PD ≥ 5 mm; mininum 16 teeth in both jaws
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Photochemotherapy; Periodontal Debridement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- laser and methilene blue (Experimental): After random allocation, all patients received full-mouth ultrasonic debridement using an ultrasonic scaler (Profi III Bios, Dabi Atlante, Ribeirão Preto, São Paulo, Brazil) for 1 hour. Specific tips were used (Perio sub, Dabi Atlante, Ribeirão Preto, São Paulo, Brazi). PDT was performed on only one side of the mouth and the initial step was subgingival irrigation with 0.005% methylene blue dye. To avoid contamination of the control sites with the dye, the methylene blue was applied only inside the periodontal pockets and a high-powered suction device controlled the flow. Two minutes after applying the photosensitizer, the low power laser - AsGaAl (Photon Laser III - PL7336, DMC, São Carlos -São Paulo, Brazil) was applied (660 nm, 100 mW, 9 J, 90 seconds per site, 320 J/cm2).
  Interventions: Other: photodynamic therapy and periodontal debridement

INTERVENTIONS:
Other: photodynamic therapy and periodontal debridement — At least two teeth (one with PD ≥ 7 mm and another with PS ≥ 5 mm) were randomly assigned (by coin toss) to one of the treatments: with (test group) or without PDT (control group). After random allocation, all patients received full-mouth ultrasonic debridement using an ultrasonic scaler for 1 hour. Specific tips were used. PDT was performed on only one side of the mouth and the initial step was subgingival irrigation with 0.005% methylene blue dye. To avoid contamination of the control sites with the dye, the methylene blue was applied only inside the periodontal pockets and a high-powered suction device controlled the flow. Two minutes after applying the photosensitizer, the low power laser - AsGaAl was applied for 90 seconds.
  Other Names: debridement using an ultrasonic scaler; Specific tips were used; 0.005% methylene blue dye; low power laser - AsGaAl

SUMMARY:
Background: Photodynamic therapy (PDT) is a method of microbial reduction which can benefit periodontal treatment in areas of difficult access, such as deep pockets and furcations. The aim of this randomized controlled clinical trial was to evaluate the effects of PDT as an adjunct to full-mouth ultrasonic debridement in the treatment of severe chronic periodontitis.

Methods: Twenty-two patients with at least one pocket with probing depth (PD) ≥ 7 mm and one pocket with PD ≥ 5 mm and bleeding on probing (BOP) on each side of the mouth were included, characterizing a split mouth design. The control group underwent full-mouth ultrasonic debridement and test group received the same treatment associated with PDT. The following clinical parameters were evaluated: plaque index, gingival index, BOP, gingival recession (GR), PD, and clinical attachment level (CAL). All parameters were collected before, 1, 3 and 6 months after treatment.

DETAILED DESCRIPTION:
The present study was a randomized, blinded, controlled clinical trial, which used a split-mouth design. Prior to commencement, the study design was approved by the Ethics Committee of Bahiana School of Medicine and Public Health (12/2008). All patients were informed individually about the nature of the proposed treatment, and informed consent forms were signed.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of severe chronic periodontitis by the presence of periodontal pockets with clinical attachment loss (CAL) ≥ 5 mm, bleeding on probing (BOP) and radiographic bone loss12;
* minimum of 2 teeth with probing depth (PD) ≥ 7 mm and 2 other teeth with PD ≥ 5 mm, all with BOP and located on opposite sides of the mouth; and
* ≥ 16 teeth in both jaws (wisdom teeth excluded).

Exclusion Criteria:

* periapical alterations on qualifying teeth,
* systemic diseases that require prophylaxis antibiotic coverage or that could influence progression and response to treatment
* periodontal treatment in the preceding 6 months,
* consumption of antibiotic, anti-inflammatory, anticonvulsant, immunosuppressant or calcium channel blocker within the past 3 months; pregnancy;
* orthodontic therapy,
* smoking and
* cardiac pace-makers users

Ages: 31 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in clinical attachment level | 1,3, 6 months
  Photodynamic therapy associated with full-mouth ultrasonic debridement in the treatment of severe chronic periodontitis: a randomized-controlled clinical trial Running title: Photodynamic therapy associated with periodontal debridement
Photodynamic therapy and periodontitis chronic severe | 1 and 3 months
  An improvement in BOP, PD and CAL was observed after treatment, in both groups, but without difference them.

SECONDARY OUTCOMES:
changes in clinical attachment level Running title: Photodynamic therapy associated with periodontal debridement Photodynamic th | 1,3, 6 months
  An improvement in BOP, PD and CAL was observed after treatment, in both groups, but without difference them. After 6 months, PD decreased from 5.11 ± 0.56 mm to 2.83 ± 0.47 mm in test group (p<0.05) and from 5.15 ± 0.46 mm to 2.83 ± 0.40 mm in control group (p<0.05). The CAL changed, after 6 months, from 5.49 ± 0.76 mm to 3.41 ± 0.84 mm in th test group (p<0.05) and from 5.53 ± 0.54 to 3.39 ± 0.51 mm in control group (p<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Maybel Balata, Master, Principal Investigator — Master and Especialist in Periodontics of Bahiana School of Medicine and Public Health, Salvador, BA, Brazil.